CLINICAL TRIAL: NCT02052336
Title: An Open-label, Randomized, 6-Sequence, 3-Period Crossover Study to Evaluate a Pharmacokinetic Drug Interaction Between CJ-12420 and Clarithromycin in Healthy Male Subjects
Brief Title: Drug-Drug Interaction Study Between CJ-12420 and Clarithromycin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_APA_103
Record Dates: First submitted 2014-01-07; First posted 2014-02-03 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Drug-Drug interaction; Pharmacokinetics
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CJ-12420 200 mg + Clarithromycin 500mg (Experimental): CJ-12420 200mg QD for 5 days + Clarithromycin 500mg BID for 5 days
  Interventions: Drug: CJ-12420 200mg; Drug: Clarithromycin 500mg
- CJ-12420 200mg (Active Comparator): CJ-12420 200mg QD for 5 days
  Interventions: Drug: CJ-12420 200mg + Clarithromycin 500mg; Drug: Clarithromycin 500mg
- Clarithromycin 500mg (Active Comparator): Clarithromycin 500mg BID for 5 days
  Interventions: Drug: CJ-12420 200mg + Clarithromycin 500mg; Drug: CJ-12420 200mg

INTERVENTIONS:
Drug: CJ-12420 200mg + Clarithromycin 500mg — To assess the effect of the coadministration of multiple dose of CJ-12420 and clarithromycin on the pharmacokinetics (PK) of CJ-12420 or clarithromycin.
  Other Names: CJ-12420 200mg for 5 days + Clarithromycin 500mg for 5 days
  Arms: CJ-12420 200mg; Clarithromycin 500mg
Drug: CJ-12420 200mg — To assess the effect of the coadministration of multiple dose of CJ-12420 and clarithromycin on the pharmacokinetics (PK) of CJ-12420 or clarithromycin.
  Other Names: CJ-12420 200mg for 5 days
  Arms: CJ-12420 200 mg + Clarithromycin 500mg; Clarithromycin 500mg
Drug: Clarithromycin 500mg — To assess the effect of the coadministration of multiple dose of CJ-12420 and clarithromycin on the pharmacokinetics (PK) of CJ-12420 or clarithromycin.
  Other Names: Clarithromycin 500mg for 5 days
  Arms: CJ-12420 200 mg + Clarithromycin 500mg; CJ-12420 200mg

SUMMARY:
Primary Objective: To assess the effect of the coadministration of multiple dose of CJ-12420 and clarithromycin on the pharmacokinetics (PK) of CJ-12420 or clarithromycin.

Secondary Objective(s): To assess the safety of the coadministration of multiple dose of CJ-12420 and clarithromycin in healthy subjects

DETAILED DESCRIPTION:
An open-label, randomized, 6-sequence, 3-period, 3-treatment crossover design

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers in the age between 19 and 45 years old
* Body mass index(BMI) in the range of 19 to 28 kg/m2
* Understand the requirement of the study and voluntarily consent to paticipate in the study

Exclusion Criteria:

* History of clinically significant medical history or disease (hepatic, kidney, gastrointestinal,respiratory, musculoskeletal, endocrine,neuro-psychiatric, haemato-oncologic,urinary tract, cardiac arrhythmia and cardiovascular system) judged by investigator.
* Clinically significant abnormal laboratory results within at least 28 days prior to the first day of drug administration. AST or ALT > 1.25 times of upper limit value Total bilirubin > 1.5 times of upper limit value estimated GFR :less than 80 mL/min
* Clinically significant abnormal ECG results within at least 28 days prior to the first day of drug administration PR ≥ 210 msec QRS ≥ 120 msec QT ≥ 500 msec QTcF ≥ 500 msec
* Clinically significant hypersensitivity reaction against investigational drug or other drugs
* history of drug abuse or "positive" results from drug screening test.
* Take medicine such as prescription medicine or herbal medicine, over-the-counter drug, vitamin supplements
* Person who have intake history of food or drug which can affect drug absorption, drug distribution, drug metabolism, and drug excretion and bowel activity
* Volunteer have a history of donation of whole blood donation, apheresis, transfusion
* Volunteer a heavy drinker(30g/day), smoker(10 cigarettes/day), heavy caffeine consumer(400mg/day)

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The effect of the coadministration of multiple dose of CJ-12420 and clarithromycin on the pharmacokinetics (PK) of CJ-12420 or clarithromycin | Blood sampling during 12 or 24hrs after administration
  Cmax, Cmin, Tmax, AUC(tau), CL/F, T1/2

SECONDARY OUTCOMES:
The safety of the coadministration of multiple dose of CJ-12420 and clarithromycin in healthy subjects | 6 days after last visit
  Safety and tolerability parameters will include laboratory (haematology, clinical chemistry, urinalysis, 12-lead ECG) values at Screening, Day-1 and Day 6 at each period and Follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Inje university college of medicine Busan Paik Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oh M, Lee H, Kim S, Kim B, Song GS, Shin JG, Ghim JL. Evaluation of pharmacokinetic drug-drug interaction between tegoprazan and clarithromycin in healthy subjects. Transl Clin Pharmacol. 2023 Jun;31(2):114-123. doi: 10.12793/tcp.2023.31.e11. Epub 2023 Jun 27. PMID 37440779